CLINICAL TRIAL: NCT05408429
Title: A PHASE 3, RANDOMIZED, PARTIALLY DOUBLE-BLIND TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN HEALTHY TODDLERS 12 THROUGH 23 MONTHS OF AGE WITH 2 PRIOR INFANT DOSES OF PREVENAR 13
Brief Title: Safety and Immunogenicity of 20vPnC in Toddlers With 2 Prior Doses of Prevenar 13
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B7471027; 2021-006624-41 (EudraCT Number)
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is partially masked. Participants randomized to receive 2 doses of 20vPnC will not have treatment masking. Participants randomized to receive 1 dose of 20vPnC or 13vPnC will have treatment masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2-Dose 20vPnC Group (Experimental): Pneumococcal conjugate vaccine (2 doses approximately 2 months apart)
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine
- 1-Dose 20vPnC Group (Experimental): Pneumococcal conjugate vaccine
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine
- 13vPnC Group (Active Comparator): Pneumococcal conjugate vaccine
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 20-valent pneumococcal conjugate vaccine — 20-valent pneumococcal conjugate vaccine
  Arms: 1-Dose 20vPnC Group; 2-Dose 20vPnC Group
Biological: 13-valent pneumococcal conjugate vaccine — 13-valent pneumococcal conjugate vaccine
  Arms: 13vPnC Group

SUMMARY:
The purpose of this study is to understand the safety and effects of a study vaccine (20vPnC) in toddlers who had 2 prior doses of Prevnar 13.

This study is being conducted in children who:

* are between 12 to 23 months of age;
* are healthy as determined by the study doctors;
* have received 2 doses of Prevnar 13 during the first year in life.

Participants in this study will receive either 1 dose or 2 doses of the study vaccine or 1 dose of Prevnar 13 as a shot in the muscle. During the study, participants will have to come to the study clinic to receive the vaccines and have blood sample collected. The study team will work with participants' parents or legal guardians to monitor any unwanted reactions to the vaccines. Participants are expected to take part in this study for about 1 or 3 months, for 1 dose or 2 dose schedules, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male or female toddlers ≥12 to <24 months of age at the time of consent
* Healthy toddlers determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study
* 2 infant doses of Prevenar 13 prior to 12 months of age

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis)
* Major known congenital malformation or serious chronic disorder
* Other chronic medical or laboratory abnormality that may increase the risk associated with study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Previous vaccination with any investigational pneumococcal vaccine, or planned receipt through study participation

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 356 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- Hungary (8):
  - Gyerkőc- Med Szolgáltató és Kereskedelmi Betéti Társaság, Budapest
  - Lurko-Med Kft Hazi Gyermekorvosi Rendelo, Budapest
  - Elitance Duo Kft., Budapest
  - Private practice - Dr. Várhelyiné Dr. Torday Judit, Debrecen
  - Zsebibaba 2004 Bt. 8. Sz Gyermekkorzet, Eger
  - Mimiped Betéti Társaság, Győr
  - Futurenest Klinikai Kutató Kft., Miskolc
  - Papp és Társa Egészségügyi és Szolgaltató Betéti Társaság, Szigetvár
- Poland (16):
  - Rodzinne Centrum Medyczne LUBMED, Luboń, Greater Poland Voivodeship
  - MICS Centrum Medyczne Toruń, Torun, Kuyavian-Pomeranian Voivodeship
  - Przylądek Zdrowia, Krakow, Lesser Poland Voivodeship
  - SZPZOZ im. Dzieci Warszawy w Dziekanowie Lesnym, Łomianki, Masovian Voivodeship
  - IN-VIVO Bydgoszcz, Bydgoszcz
  - SZPZOZ im. Dzieci Warszawy w Dziekanowie Lesnym, Dziekanów Leśny
  - Pro Familia Altera Sp. z o.o., Katowice
  - NZOZ Vita Longa Sp. z o.o., Katowice
  - Przylądek Zdrowia, Krakow
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow
  - Specjalistyczny Zespol Opieki Zdrowotnej nad Matka i Dzieckiem w Poznaniu, Poznan
  - Specjalistyczny Zespół Opieki Zdrowotnej nad Matką i Dzieckiem w Poznaniu, Poznan
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - MICS Centrum Medyczne Toruń, Torun
  - Szpital Bielanski im. Ks. Jerzego Popieluszki SPZOZ w Warszawie, Warsaw
  - Uniwersytecki Szpital Kliniczny im. J. Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Spain (18):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [LA Coruña]
  - Hospital Germans Trias i Pujol, Badalona, Barcelona [barcelona]
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona [barcelona]
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona
  - EAP Osona Sud - Alt Congost S.L.P, Centelles, Catalunya [cataluña]
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela, LA Coruña
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, LA Coruña
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte, Madrid
  - Hospital Universitario HM Puerta del Sur, Madrid, Madrid, Comunidad de
  - Grupo Pediatrico Uncibay, Málaga, Málaga
  - Hospital de Nens de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Grupo Pediatrico Uncibay, Málaga
  - Instituto Hispalense de Pediatria, Seville

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Martinon-Torres F, Martinez SN, Kline MJ, Drozd J, Trammel J, Peng Y, Giardina PC, Gruber WC, Watson W, Bickham K, Tamimi N. A phase 3 study of 20-valent pneumococcal conjugate vaccine in healthy toddlers previously vaccinated in infancy with 13-valent pneumococcal conjugate vaccine. Vaccine. 2025 Apr 19;53:126931. doi: 10.1016/j.vaccine.2025.126931. Epub 2025 Mar 12. PMID 40081152
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471027

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants included in this study were toddlers greater than or equal to (>=) 12 to less than (<) 24 months of age who had received 2 doses of 13-valent pneumococcal conjugate vaccine (13vPnC) (Prevenar 13) in infancy (prior to 12 months of age).
Pre-assignment Details: A total of 356 participants were enrolled and randomized to receive either 2 dose of 20-valent pneumococcal conjugate vaccine (20vPnC), 1 dose of 20vPnC or 1 dose of 13vPnC.
Groups:
- 2-Dose 20vPnC: Toddlers >=12 to <24 months of age were randomized to receive 2 doses of 0.5 milliliter (mL) 20vPnC intramuscularly. Dose 1 was administered at Day 1 (Dose 1 Visit) and Dose 2 was administered 56 to 70 days later (Dose 2 Visit).
- 1-Dose 20vPnC: Toddlers >=12 to <24 months of age were randomized to receive 1 dose of 0.5 mL 20vPnC intramuscularly on Day 1 (Dose 1 Visit).
- 13vPnC Control: Toddlers >=12 to <24 months of age were randomized to receive 1 dose of 0.5 mL 13vPnC intramuscularly on Day 1 (Dose 1 Visit).
Period: Overall Study
Arm/Group | 2-Dose 20vPnC | 1-Dose 20vPnC | 13vPnC Control
Started | 121 | 118 | 117
Completed | 115 | 117 | 116
Not Completed | 6 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who receive at least 1 dose of the study intervention and have safety data reported after any dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2-Dose 20vPnC | 1-Dose 20vPnC | 13vPnC Control | Total
Number analyzed (Participants) | 121 | 118 | 117 | 356
Age, Continuous [Mean (Standard Deviation); unit: months] | 12.5 (1.21) | 12.6 (1.52) | 12.7 (1.85) | 12.6 (1.54)
Age, Customized [Count of Participants; unit: Participants]
  Infants and toddlers (28 days-23 months) | 121 | 118 | 117 | 356
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 47 | 57 | 164
  Male | 61 | 71 | 60 | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 36 | 32 | 102
  Not Hispanic or Latino | 86 | 82 | 85 | 253
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 120 | 117 | 113 | 350
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Last Vaccination
Description: Local reactions included redness, swelling, and pain at the injection site, recorded by parents/legal guardians of participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device (caliper) units. 1 measuring device unit = 0.5 centimeter (cm). Redness and swelling were graded as mild (greater than [>] 0 to 2.0 cm), moderate (>2.0 to 7.0 cm) and severe (>7.0 cm). Pain at injection site was graded as mild (hurt if gently touched example, whimpered, winced, protested, or withdrew), moderate (hurt if gently touched, with crying), and severe (caused limitation of limb movement). 95 percent (%) confidence interval (CI) was based on Clopper and Pearson method.
Time Frame: Within 7 days after last vaccination (for reporting arm 2-Dose 20vPnC last vaccination was Dose 2 and for 1-dose 20vPnC and 13vPnC Control it was Dose 1)
Population: Safety analysis set included all participants who received at least 1 dose of 20vPnC or 13vPnC and had safety data reported after any dose. Here, "Number of Participants Analyzed" signifies the number of participants with any e-diary data reported after the last vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose 20vPnC | 1-Dose 20vPnC | 13vPnC Control
Number analyzed (Participants) | 114 | 118 | 117
Percentage of participants
  Redness: Any | 26.3 (18.5) [18.5 to 35.4] | 29.7 (21.6) [21.6 to 38.8] | 32.5 (24.1) [24.1 to 41.8]
  Redness: Mild | 13.2 (7.6) [7.6 to 20.8] | 18.6 (12.1) [12.1 to 26.9] | 17.9 (11.5) [11.5 to 26.1]
  Redness: Moderate | 12.3 (6.9) [6.9 to 19.7] | 11.0 (6.0) [6.0 to 18.1] | 14.5 (8.7) [8.7 to 22.2]
  Redness: Severe | 0.9 (0.0) [0.0 to 4.8] | 0 (0.0) [0.0 to 3.1] | 0 (0.0) [0.0 to 3.1]
  Swelling: Any | 23.7 (16.2) [16.2 to 32.6] | 21.2 (14.2) [14.2 to 29.7] | 25.6 (18.0) [18.0 to 34.5]
  Swelling: Mild | 14.0 (8.2) [8.2 to 21.8] | 12.7 (7.3) [7.3 to 20.1] | 16.2 (10.1) [10.1 to 24.2]
  Swelling: Moderate | 8.8 (4.3) [4.3 to 15.5] | 8.5 (4.1) [4.1 to 15.0] | 9.4 (4.8) [4.8 to 16.2]
  Swelling: Severe | 0.9 (0.0) [0.0 to 4.8] | 0 (0.0) [0.0 to 3.1] | 0 (0.0) [0.0 to 3.1]
  Pain at Injection Site: Any | 29.8 (21.6) [21.6 to 39.1] | 28.8 (20.8) [20.8 to 37.9] | 31.6 (23.3) [23.3 to 40.9]
  Pain at Injection Site: Mild | 17.5 (11.1) [11.1 to 25.8] | 17.8 (11.4) [11.4 to 25.9] | 26.5 (18.8) [18.8 to 35.5]
  Pain at Injection Site: Moderate | 12.3 (6.9) [6.9 to 19.7] | 11.0 (6.0) [6.0 to 18.1] | 5.1 (1.9) [1.9 to 10.8]
  Pain at Injection Site: Severe | 0 (0.0) [0.0 to 3.2] | 0 (0.0) [0.0 to 3.1] | 0 (0.0) [0.0 to 3.1]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Last Vaccination
Description: Systemic events included fever, decreased appetite, drowsiness/increased sleep and irritability, recorded by parents/legal guardians of participants using an e-diary. Fever: temperature >=38.0 degree Celsius (C) and categorized as >=38.0 to 38.4 degree C,>38.4 to 38.9 degree C,>38.9 to 40.0 degree C and >40.0 degree C. Decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased/prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity). Irritability was graded as mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted). 95% CI was based on Clopper & Pearson method.
Time Frame: as for outcome 1
Population: Safety analysis set included all participants who received at least 1 dose of 20vPnC or 13vPnC and had safety data assessed after any dose. Here, "Number of Participants Analyzed" signifies number of participants with any e-diary data reported after the last vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose 20vPnC | 1-Dose 20vPnC | 13vPnC Control
Number analyzed (Participants) | 114 | 118 | 117
Percentage of participants
  Fever: >=38.0 degrees C | 9.6 (4.9) [4.9 to 16.6] | 15.3 (9.3) [9.3 to 23.0] | 15.4 (9.4) [9.4 to 23.2]
  Fever: >38.0 degrees C to 38.4 degrees C | 3.5 (1.0) [1.0 to 8.7] | 6.8 (3.0) [3.0 to 12.9] | 10.3 (5.4) [5.4 to 17.2]
  Fever: >38.4 degrees C to 38.9 degrees C | 4.4 (1.4) [1.4 to 9.9] | 3.4 (0.9) [0.9 to 8.5] | 2.6 (0.5) [0.5 to 7.3]
  Fever: >38.9 degrees C to 40.0 degrees C | 1.8 (0.2) [0.2 to 6.2] | 5.1 (1.9) [1.9 to 10.7] | 2.6 (0.5) [0.5 to 7.3]
  Fever: >40.0 degrees C | 0 (0.0) [0.0 to 3.2] | 0 (0.0) [0.0 to 3.1] | 0 (0.0) [0.0 to 3.1]
  Decreased appetite: Any | 25.4 (17.7) [17.7 to 34.4] | 33.1 (24.7) [24.7 to 42.3] | 26.5 (18.8) [18.8 to 35.5]
  Decreased appetite: Mild | 14.9 (8.9) [8.9 to 22.8] | 15.3 (9.3) [9.3 to 23.0] | 12.0 (6.7) [6.7 to 19.3]
  Decreased appetite: Moderate | 10.5 (5.6) [5.6 to 17.7] | 14.4 (8.6) [8.6 to 22.1] | 13.7 (8.0) [8.0 to 21.3]
  Decreased appetite: Severe | 0 (0.0) [0.0 to 3.2] | 3.4 (0.9) [0.9 to 8.5] | 0.9 (0.0) [0.0 to 4.7]
  Drowsiness/increased sleep: Any | 23.7 (16.2) [16.2 to 32.6] | 32.2 (23.9) [23.9 to 41.4] | 31.6 (23.3) [23.3 to 40.9]
  Drowsiness/increased sleep: Mild | 18.4 (11.8) [11.8 to 26.8] | 25.4 (17.9) [17.9 to 34.3] | 21.4 (14.3) [14.3 to 29.9]
  Drowsiness/increased sleep: Moderate | 5.3 (2.0) [2.0 to 11.1] | 5.9 (2.4) [2.4 to 11.8] | 10.3 (5.4) [5.4 to 17.2]
  Drowsiness/increased sleep: Severe | 0 (0.0) [0.0 to 3.2] | 0.8 (0.0) [0.0 to 4.6] | 0 (0.0) [0.0 to 3.1]
  Irritability: Any | 55.3 (45.7) [45.7 to 64.6] | 50.8 (41.5) [41.5 to 60.2] | 46.2 (36.9) [36.9 to 55.6]
  Irritability: Mild | 24.6 (17.0) [17.0 to 33.5] | 15.3 (9.3) [9.3 to 23.0] | 16.2 (10.1) [10.1 to 24.2]
  Irritability: Moderate | 29.8 (21.6) [21.6 to 39.1] | 32.2 (23.9) [23.9 to 41.4] | 29.9 (21.8) [21.8 to 39.1]
  Irritability: Severe | 0.9 (0.0) [0.0 to 4.8] | 3.4 (0.9) [0.9 to 8.5] | 0 (0.0) [0.0 to 3.1]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Last Vaccination to 1 Month After Last Vaccination
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. 95% CI was based on the Clopper and Pearson method. AEs reported in this endpoint excluded local reactions and systemic events collected from an e-diary.
Time Frame: From last vaccination to 1 Month after last vaccination (for reporting arm 2-Dose 20vPnC last vaccination was Dose 2 and for 1-dose 20vPnC and 13vPnC Control it was Dose 1)
Population: Safety analysis set included all participants who received at least 1 dose of 20vPnC or 13vPnC and had safety data assessed after any dose. Here, "Number of Participants Analyzed" signifies the number of participants in the specified group who received the last vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose 20vPnC | 1-Dose 20vPnC | 13vPnC Control
Number analyzed (Participants) | 116 | 118 | 117
Percentage of participants | 22.4 (15.2) [15.2 to 31.1] | 24.6 (17.1) [17.1 to 33.4] | 25.6 (18.0) [18.0 to 34.5]

4. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) From Last Vaccination to 1 Month After Last Vaccination
Description: A SAE was any untoward medical occurrence that: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/ incapacity; was a congenital anomaly/birth defect; was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic, was considered serious and other important medical events. 95% CI was based on the Clopper and Pearson method.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose 20vPnC | 1-Dose 20vPnC | 13vPnC Control
Number analyzed (Participants) | 116 | 118 | 117
Percentage of participants | 0.9 (0.0) [0.0 to 4.7] | 0.8 (0.0) [0.0 to 4.6] | 0.9 (0.0) [0.0 to 4.7]

5. Primary Outcome: Percentage of Participants With Predefined Serotype-Specific Immunoglobulin G (IgG) Concentrations for the 7 Additional Serotypes 1 Month After Last Vaccination
Description: Pneumococcal serotype-specific IgG concentrations were measured for serum samples for 7 additional serotypes: 8, 10A, 11A, 12F, 15B, 22F, 33F. The predefined level was 0.35 microgram per milliliter (mcg/mL) for all 7 additional serotypes. 95% CI was based on the Clopper and Pearson method.
Time Frame: 1 Month after last vaccination (for reporting arm 2-Dose 20vPnC last vaccination was Dose 2 and for 1-dose 20vPnC and 13vPnC Control it was Dose 1)
Population: Evaluable immunogenicity population (EIP) included all participants who were eligible, received vaccinations to which they were randomized, had at least 1 valid immunogenicity result from 1 month after the last assigned vaccination collected within 27 to 56 days after the dose, had no other major protocol deviations as determined by clinician. "Number of Participants analyzed"= participants in EIP. "Number analyzed"= participants with valid IgG results for specified serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose 20vPnC | 1-Dose 20vPnC | 13vPnC Control
Number analyzed (Participants) | 102 | 108 | 108
Percentage of participants
  Serotype 8: number analyzed (Participants) | 102 | 108 | 107
  Serotype 8 | 100.0 [96.4 to 100.0] | 98.1 [93.5 to 99.8] | 8.4 [3.9 to 15.4]
  Serotype 10A | 99.0 [94.7 to 100.0] | 87.0 [79.2 to 92.7] | 1.9 [0.2 to 6.5]
  Serotype 11A | 99.0 [94.7 to 100.0] | 96.3 [90.8 to 99.0] | 13.0 [7.3 to 20.8]
  Serotype 12F | 91.2 [83.9 to 95.9] | 54.6 [44.8 to 64.2] | 0.0 [0.0 to 3.4]
  Serotype 15B | 100.0 [96.4 to 100.0] | 75.9 [66.7 to 83.6] | 6.5 [2.6 to 12.9]
  Serotype 22F | 100.0 [96.4 to 100.0] | 94.4 [88.3 to 97.9] | 2.8 [0.6 to 7.9]
  Serotype 33F | 99.0 [94.7 to 100.0] | 83.3 [74.9 to 89.8] | 3.7 [1.0 to 9.2]

6. Secondary Outcome: Serotype-specific IgG Geometric Mean Concentrations (GMC) 1 Month After Last Vaccination
Description: Pneumococcal serotype-specific IgG concentrations were measured for serum samples for 13vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F and 7 additional serotypes: 8, 10A, 11A, 12F, 15B, 22F, 33F. Assay results below the lower limit of quantitation (LLOQ) were set to 0.5*LLOQ. GMC and corresponding 2-sided 95% CIs were calculated by exponentiating mean logarithm of concentration, corresponding 2-sided 95% CIs (based on Student's t distribution).
Time Frame: as for outcome 5
Population: EIP included all participants who were eligible, received vaccinations to which they were randomized, had at least 1 valid immunogenicity result from 1 month after the last assigned vaccination collected within 27 to 56 days after the dose, had no other major protocol deviations as determined by clinician. Here, Number of Participants Analyzed= participants in EIP. "Number Analyzed"= participants with valid IgG assay results for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 2-Dose 20vPnC | 1-Dose 20vPnC | 13vPnC Control
Number analyzed (Participants) | 102 | 108 | 108
mcg/mL
  Serotype 1 | 1.66 [1.39 to 2.00] | 2.40 [1.95 to 2.96] | 3.38 [2.82 to 4.05]
  Serotype 3 | 0.78 [0.65 to 0.93] | 0.95 [0.80 to 1.14] | 1.24 [1.06 to 1.45]
  Serotype 4 | 3.09 [2.63 to 3.63] | 4.54 [3.63 to 5.67] | 5.67 [4.81 to 6.70]
  Serotype 5 | 1.61 [1.36 to 1.92] | 2.03 [1.64 to 2.51] | 2.46 [2.04 to 2.95]
  Serotype 6A | 8.55 [7.25 to 10.07] | 12.45 [10.16 to 15.27] | 16.28 [13.48 to 19.66]
  Serotype 6B: number analyzed (Participants) | 102 | 108 | 107
  Serotype 6B | 5.17 [4.25 to 6.29] | 4.87 [3.60 to 6.60] | 6.64 [5.19 to 8.52]
  Serotype 7F | 4.78 [4.15 to 5.49] | 4.41 [3.81 to 5.10] | 6.32 [5.49 to 7.28]
  Serotype 9V | 3.44 [2.96 to 3.99] | 3.94 [3.29 to 4.71] | 5.36 [4.55 to 6.31]
  Serotype 14 | 5.58 [4.66 to 6.68] | 7.37 [5.85 to 9.29] | 8.64 [7.01 to 10.64]
  Serotype 18C | 2.84 [2.39 to 3.39] | 3.13 [2.62 to 3.74] | 3.78 [3.14 to 4.54]
  Serotype 19A | 3.31 [2.80 to 3.90] | 6.36 [5.22 to 7.74] | 6.89 [5.76 to 8.23]
  Serotype 19F: number analyzed (Participants) | 102 | 107 | 108
  Serotype 19F | 5.25 [4.38 to 6.28] | 8.78 [7.04 to 10.94] | 10.09 [8.33 to 12.22]
  Serotype 23F | 5.06 [4.23 to 6.05] | 4.45 [3.58 to 5.53] | 6.32 [5.07 to 7.89]
  Serotype 8: number analyzed (Participants) | 102 | 108 | 107
  Serotype 8 | 10.16 [8.75 to 11.79] | 7.56 [6.22 to 9.19] | 0.05 [0.04 to 0.07]
  Serotype 10A | 6.54 [5.17 to 8.28] | 1.32 [0.98 to 1.76] | 0.01 [0.01 to 0.02]
  Serotype 11A | 4.83 [4.11 to 5.68] | 2.72 [2.17 to 3.41] | 0.03 [0.02 to 0.04]
  Serotype 12F | 1.72 [1.40 to 2.12] | 0.33 [0.25 to 0.45] | 0.01 [0.01 to 0.01]
  Serotype 15B | 11.21 [9.39 to 13.38] | 0.95 [0.74 to 1.21] | 0.03 [0.02 to 0.04]
  Serotype 22F | 15.45 [13.24 to 18.03] | 8.66 [6.27 to 11.98] | 0.01 [0.00 to 0.01]
  Serotype 33F | 4.94 [4.04 to 6.03] | 1.68 [1.21 to 2.34] | 0.02 [0.01 to 0.02]

7. Secondary Outcome: Percentage of Participants With Predefined IgG Concentrations for the 13 Matched Serotypes 1 Month After Last Vaccination
Description: Pneumococcal serotype-specific IgG concentrations were measured for serum samples for 13vPnC serotypes:1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C,19A,19F, 23F. Predefined level was 0.35 mcg/mL for all 13vPnC serotypes except serotypes 5, 6B, and 19A, which had predefined levels of 0.23, 0.10, and 0.12 mcg/mL, respectively. 95% CI was based on the Clopper and Pearson method.
Time Frame: as for outcome 5
Population: EIP included all participants who were eligible, received vaccinations to which they were randomized, had at least 1 valid immunogenicity result from 1 month after last assigned vaccination collected within 27 to 56 days after dose, had no other major protocol deviations. Here, Number of Participants Analyzed= participants in EIP. "Number Analyzed"=participants with valid IgG results for specified serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2-Dose 20vPnC | 1-Dose 20vPnC | 13vPnC Control
Number analyzed (Participants) | 102 | 108 | 108
Percentage of participants
  Serotype 1 | 94.1 [87.6 to 97.8] | 94.4 [88.3 to 97.9] | 98.1 [93.5 to 99.8]
  Serotype 3 | 88.2 [80.4 to 93.8] | 87.0 [79.2 to 92.7] | 93.5 [87.1 to 97.4]
  Serotype 4 | 98.0 [93.1 to 99.8] | 99.1 [94.9 to 100.0] | 100.0 [96.6 to 100.0]
  Serotype 5 | 97.1 [91.6 to 99.4] | 96.3 [90.8 to 99.0] | 100.0 [96.6 to 100.0]
  Serotype 6A | 100.0 [96.4 to 100.0] | 99.1 [94.9 to 100.0] | 99.1 [94.9 to 100.0]
  Serotype 6B: number analyzed (Participants) | 102 | 108 | 107
  Serotype 6B | 100.0 [96.4 to 100.0] | 98.1 [93.5 to 99.8] | 100.0 [96.6 to 100.0]
  Serotype 7F | 100.0 [96.4 to 100.0] | 100.0 [96.6 to 100.0] | 100.0 [96.6 to 100.0]
  Serotype 9V | 100.0 [96.4 to 100.0] | 99.1 [94.9 to 100.0] | 100.0 [96.6 to 100.0]
  Serotype 14 | 100.0 [96.4 to 100.0] | 99.1 [94.9 to 100.0] | 99.1 [94.9 to 100.0]
  Serotype 18C | 100.0 [96.4 to 100.0] | 98.1 [93.5 to 99.8] | 99.1 [94.9 to 100.0]
  Serotype 19A | 100.0 [96.4 to 100.0] | 100.0 [96.6 to 100.0] | 100.0 [96.6 to 100.0]
  Serotype 19F: number analyzed (Participants) | 102 | 107 | 108
  Serotype 19F | 100.0 [96.4 to 100.0] | 99.1 [94.9 to 100.0] | 100.0 [96.6 to 100.0]
  Serotype 23F | 99.0 [94.7 to 100.0] | 99.1 [94.9 to 100.0] | 97.2 [92.1 to 99.4]

8. Secondary Outcome: Serotype-Specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) 1 Month After Last Vaccination
Description: OPA titers for the 20 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F, and 33F) were determined in randomly selected subsets of participants at 1 month after last vaccination received. OPA titers below the LLOQ were set to 0.5*LLOQ. GMTs and 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs based on the Student's t distribution.
Time Frame: as for outcome 5
Population: EIP: eligible participants who received vaccinations as randomized, had at least 1 valid immunogenicity result from 1 month after last dose collected within 27-56 days after dose, had no other major protocol deviation. Number of Participants Analyzed = participants in EIP. OPA titers from randomly selected participants were measured for a subset of the 20 serotypes. Number Analyzed = participants with valid OPA assay result for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 2-Dose 20vPnC | 1-Dose 20vPnC | 13vPnC Control
Number analyzed (Participants) | 102 | 108 | 108
Titers
  Serotype 1: number analyzed (Participants) | 25 | 32 | 34
  Serotype 1 | 46 [26 to 82] | 79 [47 to 133] | 105 [68 to 162]
  Serotype 3: number analyzed (Participants) | 25 | 33 | 32
  Serotype 3 | 131 [106 to 163] | 101 [72 to 142] | 128 [93 to 176]
  Serotype 4: number analyzed (Participants) | 30 | 31 | 32
  Serotype 4 | 348 [178 to 681] | 425 [213 to 845] | 541 [298 to 984]
  Serotype 5: number analyzed (Participants) | 26 | 33 | 34
  Serotype 5 | 46 [30 to 69] | 77 [52 to 114] | 73 [52 to 104]
  Serotype 6A: number analyzed (Participants) | 25 | 33 | 34
  Serotype 6A | 1470 [1030 to 2096] | 1156 [768 to 1739] | 1796 [1286 to 2508]
  Serotype 6B: number analyzed (Participants) | 26 | 32 | 33
  Serotype 6B | 698 [437 to 1114] | 452 [275 to 743] | 790 [459 to 1357]
  Serotype 7F: number analyzed (Participants) | 26 | 30 | 29
  Serotype 7F | 1415 [844 to 2371] | 1212 [755 to 1945] | 1367 [790 to 2365]
  Serotype 9V: number analyzed (Participants) | 28 | 30 | 31
  Serotype 9V | 1719 [928 to 3185] | 1792 [1015 to 3166] | 1930 [1048 to 3556]
  Serotype 14: number analyzed (Participants) | 23 | 30 | 32
  Serotype 14 | 844 [474 to 1501] | 1245 [837 to 1852] | 558 [308 to 1011]
  Serotype 18C: number analyzed (Participants) | 29 | 31 | 31
  Serotype 18C | 1861 [1115 to 3106] | 1047 [583 to 1882] | 1149 [684 to 1930]
  Serotype 19A: number analyzed (Participants) | 26 | 30 | 31
  Serotype 19A | 512 [283 to 925] | 731 [401 to 1332] | 973 [560 to 1688]
  Serotype 19F: number analyzed (Participants) | 25 | 32 | 34
  Serotype 19F | 473 [257 to 873] | 470 [285 to 775] | 595 [363 to 975]
  Serotype 23F: number analyzed (Participants) | 28 | 30 | 32
  Serotype 23F | 727 [382 to 1382] | 472 [255 to 876] | 721 [439 to 1186]
  Serotype 8: number analyzed (Participants) | 33 | 32 | 33
  Serotype 8 | 3446 [2282 to 5203] | 1609 [989 to 2617] | 76 [42 to 137]
  Serotype 10A: number analyzed (Participants) | 36 | 33 | 32
  Serotype 10A | 6783 [4555 to 10100] | 2506 [1425 to 4407] | 64 [40 to 104]
  Serotype 11A: number analyzed (Participants) | 36 | 30 | 30
  Serotype 11A | 3827 [1975 to 7414] | 3416 [1523 to 7665] | 235 [99 to 562]
  Serotype 12F: number analyzed (Participants) | 32 | 31 | 32
  Serotype 12F | 17398 [11121 to 27218] | 7346 [3895 to 13855] | 64 [34 to 122]
  Serotype 15B: number analyzed (Participants) | 35 | 29 | 34
  Serotype 15B | 10024 [6200 to 16206] | 3898 [1867 to 8136] | 58 [24 to 143]
  Serotype 22F: number analyzed (Participants) | 35 | 31 | 33
  Serotype 22F | 11820 [7993 to 17480] | 6117 [3289 to 11376] | 28 [13 to 61]
  Serotype 33F: number analyzed (Participants) | 33 | 32 | 32
  Serotype 33F | 43671 [28126 to 67809] | 15355 [9431 to 24998] | 694 [432 to 1115]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events (systematic assessment): Within 7 days after Dose 1 and 2; All-cause mortality, SAEs and non-SAEs (non-systematic assessment): from Dose 1 to 1 month after Dose 1 (1-dose groups) or Dose 2 (2-dose group)
Description: Same event may appear as both SAE and non-SAE. But what is presented are distinct events. Event may be classified as serious in 1 participant and non-serious in another, or 1 participant may have experienced both during study. Safety analysis set analyzed. Results are summarized by: 2-Dose 20vPnC Dose1 to Dose 2, 2-Dose 20vPnC (Dose 2 to 1 month after Dose 2), 1-Dose 20vPnC and 13vPnC Control.
Groups:
- 2-Dose 20vPnC (Dose 1 to Dose 2): Toddlers >=12 to <24 months of age were randomized to receive 2 doses of 0.5 mL 20vPnC intramuscularly. Dose 1 was administered at Day 1 (Dose 1 Visit) and Dose 2 was administered 56 to 70 days later (Dose 2 Visit). This arm reports data from Dose 1 to Dose 2.
- 2-Dose 20vPnC (Dose 2 to 1 Month After Dose 2): Toddlers >=12 to <24 months of age were randomized to receive 2 doses of 0.5 mL 20vPnC intramuscularly. Dose 1 was administered at Day 1 (Dose 1 Visit) and Dose 2 was administered 56 to 70 days later (Dose 2 Visit). This arm reports data From Dose 2 to 1 month after Dose 2.
- 1-Dose 20vPnC (Dose 1 to 1 Month After Dose 1); 13vPnC Control (Dose 1 to 1 Month After Dose 1): Toddlers >=12 to <24 months of age were randomized to receive 1 dose of 0.5 mL 20vPnC intramuscularly on Day 1 (Dose 1 Visit). This arm reports data from dose 1 to 1 month after Dose 1.
Arm/Group | 2-Dose 20vPnC (Dose 1 to Dose 2) | 2-Dose 20vPnC (Dose 2 to 1 Month After Dose 2) | 1-Dose 20vPnC (Dose 1 to 1 Month After Dose 1) | 13vPnC Control (Dose 1 to 1 Month After Dose 1)
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/116 | 0/118 | 0/117
Serious Adverse Events (participants affected / at risk) | 4/121 | 1/116 | 1/118 | 1/117
Other Adverse Events (participants affected / at risk) | 93/121 | 91/116 | 90/118 | 98/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-Dose 20vPnC (Dose 1 to Dose 2) (N=121) | 2-Dose 20vPnC (Dose 2 to 1 Month After Dose 2) (N=116) | 1-Dose 20vPnC (Dose 1 to 1 Month After Dose 1) (N=118) | 13vPnC Control (Dose 1 to 1 Month After Dose 1) (N=117)
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2-Dose 20vPnC (Dose 1 to Dose 2) (N=121) | 2-Dose 20vPnC (Dose 2 to 1 Month After Dose 2) (N=116) | 1-Dose 20vPnC (Dose 1 to 1 Month After Dose 1) (N=118) | 13vPnC Control (Dose 1 to 1 Month After Dose 1) (N=117)
Hypersomnia (INCREASED SLEEP) (Nervous system disorders) | 39 | 27 | 38 | 37
Decreased appetite (DECREASED APPETITE) (Metabolism and nutrition disorders) | 37 | 29 | 39 | 31
Upper respiratory tract infection (Infections and infestations) | 18 | 9 | 13 | 9
Injection site erythema (REDNESS) (General disorders) | 40 | 30 | 35 | 38
Injection site pain (PAIN) (General disorders) | 33 | 34 | 34 | 37
Injection site swelling (SWELLING) (General disorders) | 27 | 27 | 25 | 30
Pyrexia (FEVER) (General disorders) | 20 | 11 | 18 | 18
Irritability (Psychiatric disorders) | 70 | 63 | 60 | 54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT05408429/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT05408429/SAP_001.pdf